CLINICAL TRIAL: NCT07197541
Title: A Self-controlled Study of Bleomycin and Pingyangmycin Injection in the Treatment of Plantar Warts
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0001
Record Dates: First submitted 2024-10-06; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2024-10

CONDITIONS: Plantar Wart
MeSH Terms: interventions — Bleomycin; bleomycetin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bleomycin group (Experimental)
  Interventions: Drug: Bleomycin Injection
- Pingyangmycin group (Experimental)
  Interventions: Drug: Pingyangmycin Injection

INTERVENTIONS:
Drug: Bleomycin Injection — Bleomycin injection treatment group: local injection treatment, once every 4 weeks.
  Arms: Bleomycin group
Drug: Pingyangmycin Injection — Pingyangmycin injection treatment group: local injection treatment, once every 4 weeks.
  Arms: Pingyangmycin group

SUMMARY:
All patients were treated as self-control. Half of the warts received bleomycin injection and the other half received pingyangmycin injection for 24 weeks. During the treatment period, before each injection, photos of the skin lesions must be taken, the diameter of the skin lesions must be measured, the DLQI(Dermatology Life Quality Index) and NRS scores(NRS scores) must be filled in, and adverse events must be recorded. Before the first treatment, HPV(Human Papilloma virus) virus typing is performed on the warts.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years old;
2. Clinical diagnosis of plantar warts;
3. The diameter of a single wart is ≥1cm, and the number is ≥2;
4. There is a history of other treatments for plantar warts within 4 weeks, including drugs and physical therapy;
5. Have a basic understanding of the purpose, effects and possible adverse reactions of the trial, and sign an informed consent form in accordance with the spirit of the Declaration of Helsinki.

Exclusion Criteria:

1. There are other local infections in the treatment area and injection is not suitable;
2. Patients allergic to lidocaine, bleomycin, and pingyangmycin;
3. Patients with other serious skin diseases, tumors or other systemic diseases;
4. Patients with infections such as tuberculosis, HIV, hepatitis B, hepatitis C;
5. Patients with a history of other treatments for plantar warts in the previous 4 weeks, including drugs and physical therapy;
6. Patients who have participated in other clinical trials in the past 3 months;
7. Pregnant women, lactating women, or patients who plan to become pregnant during the trial;
8. Those who have any history of major surgery in the previous 8 weeks or who may have surgery planned during treatment;
9. Patients with a history of mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Skin lesions completely cleared | 2026.11.1
  The patient's plantar wart lesions were completely cleared

SECONDARY OUTCOMES:
Follow up to 36 weeks with no recurrence | 2026.11.1
  There was no recurrence of plantar warts in the patient at 36 weeks of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Zhou, PhD, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No